CLINICAL TRIAL: NCT05588765
Title: Effects of Respiratory Muscle Training on Pulmonary Function of Patients With Chronic Neck Pain
Brief Title: Effects of Respiratory Muscle Training on Pulmonary Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: Riphah International University (Other)
Responsible Party: Principal Investigator, Madeeha Shafiq, Lecturer, University of Lahore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00534
Record Dates: First submitted 2022-10-03; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Chronic Neck Pain

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: Seal Envelope method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle endurance training (Experimental): Volume oriented incentive spirometer improves respiratory muscle endurance and chest expansion.
  Interventions: Other: Neck stretching exercises
- Diaphragmatic breathing exercises (Active Comparator): Improvement in diaphragm contraction, chest wall symmetry and reduce activity of accessory muscle due to diaphragmatic breathing technique causes respiratory muscle endurance to improve.
  Interventions: Other: Neck stretching exercises

INTERVENTIONS:
Other: Neck stretching exercises — Neck stretching exercises towards lateral flexion, ipsilateral flexion and rotation and towards flexion each for 30 sec and repeated 2-3 times

SUMMARY:
The study was conducted to determine the effects of respiratory muscle training on pulmonary function and musculoskeletal parameters in patients with chronic neck pain. It included 43 patients, 20-40 years old males and females having non-specific chronic neck pain for more than three months and with low maximum voluntary ventilation (MVV) values were included. Control group (n=21) received conventional physiotherapy with diaphragmatic breathing exercises and experimental group (n=23) received conventional physiotherapy with specially designed respiratory exercise protocol. It concluded that RMT in addition to conventional physiotherapy is effective to improve musculoskeletal and pulmonary parameters in CNP patients.

DETAILED DESCRIPTION:
To determine the effects of respiratory muscle training on pulmonary function and musculoskeletal parameters in patients with chronic neck pain.

Study design: A randomized controlled trial Place and Duration of Study: Riphah Rehabilitation and Research Center in Railway General Hospital and Benazir Bhutto Hospital, Rawalpindi from January 2019 to July 2019.

Methodology: 43 patients, 20-40 years old males and females having non-specific chronic neck pain for more than three months and with low maximum voluntary ventilation (MVV) values were included. Control group (n=21) received conventional physiotherapy with diaphragmatic breathing exercises and experimental group (n=23) received conventional physiotherapy with specially designed respiratory exercise protocol. They were assessed prior to, at 2nd week and after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* . Patients having non-specific chronic neck pain with or without headache for more than three months with pain complaints at least once a week 2. Males and females both of age 20 to 40 years old 3. Patients with low maximum voluntary ventilation (MVV) values i.e., less than 110 L/min in males and 80 L/min in females

Exclusion Criteria:

* Patients already participating in physiotherapy program 2. Patients with past history of

  * surgery to the cervical spine
  * traumatic cervical injuries
  * clinical abnormalities or surgeries of the thoracic cage or vertebral column
  * severe obesity (BMI>40)
  * pregnancy
  * smoking history/occupational industrial exposures
  * chronic neuro-musculoskeletal pain in any other non-related body area
  * respiratory or cardiac illness, diabetes mellitus and serious comorbidities

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pulmonary Function | Baseline and 4 weeks
  Determines possible obstruction or restriction is present in patients suspect-able to lung dysfunction
Change from baseline in Cloth tape measurement technique | Baseline and 4 weeks
  Cloth tape measurement technique is used as an outcome measure for chest expansion in management of cardio respiratory conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PHD*, Principal Investigator — Suman.sheraz@riphah.edu.pk
Locations (1):
- Suman, Islamabad, Pakistan